CLINICAL TRIAL: NCT00668174
Title: Physical Activity and Total Health Trial
Brief Title: Effect of Exercise on Sex Hormones in Postmenopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Anne McTiernan, MD, PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PATH - CA/AG69334-01A2,; IR-4290
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer Prevention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 2 (No Intervention): Control

INTERVENTIONS:
Behavioral: Exercise — Moderate intensity exercise, 5 days per week, 45 min per session, 50-70% max HR, divided into a 3-month individualized and 9-month maintenance period.
  Arms: 1

SUMMARY:
The goals of the study are to examine the effect in postmenopausal women of a one-year moderate intensity exercise intervention, as compared with a sedentary pattern (low-level stretching program), on: serum estrogens, androgens, sex hormone binding globulin, insulin, triglycerides, glucose, aromatase, FSH, LH, as well as parameters of body fat mass.

ELIGIBILITY:
Inclusion Criteria:

* Ages 55-75 years at first group meeting
* Physically able to undertake a moderate exercise program
* Sedentary activity pattern (exercising < 2 times/week for 20 minutes at a level to produce sweating)
* Postmenopausal (not experiencing menstrual periods for the previous 12 months or FSH >30 mIU/ml; for women who have had a hysterectomy, an FHS >30 mIU/ml will classify them as postmenopausal)
* Body Mass Index (BMI) greater than 25.0
* Able to follow directions and fill out questionnaires, and exercise diaries and logs in English
* Agrees to be randomly assigned to either the exercise intervention or control group
* Gives informed consent to participate in all screening and study activities
* Able to come to the FHCRC for clinic visits and classes, to the UW Medical Center for CT scans, and to the UW NETT for measurements and instruction

Exclusion Criteria:

* Plans to leave Western Washington within the follow-up period
* Using hormone replacement, tamoxifen, or oral contraceptives in past 6 months
* Currently having severe hot flashes (that might prompt participant to start hormone replacement therapy before the end of study)
* Current unstable thyroid disease or unstable dose of thyroid medications or TSH >5.0 IU/ml or <0.5 IU/ml
* Invasive cancer in the past 10 years (except nonmelanotic skin cancer)
* Any other endocrinologic abnormality
* Breast, endometrial, ovarian, or melanoma cancer or carcinoma-in-situ at any time
* Morbidly obese (BMI > 40)
* Current or planned use of corticosteroids
* Currently on or planning to enter a structured weight loss program or to take diet drugs
* Current use of certain other medications, such as any likely to interfere with adherence to an exercise program or likely to interfere with study outcomes
* Moderate to high alcohol intake (more than 2 drinks per day)
* Current smoker
* Diabetes mellitus (fasting hyperglycemia)
* Abnormal screening labs (hematocrit < 32 or > 48, white blood cells < 3.0 or > 15.0, potassium < 3.5 or > 5.0, fasting glucose > 140, creatinine > 2.0), or abnormalities on screening physical judged by study physicians to contraindicate participation in an exercise program
* Contraindications for entry into a training program118 including: unstable angina, uncontrolled hypertension (systolic > 200, diastolic > 100), orthostatic hypotension (> 20), moderate/severe aortic stenosis, uncontrolled arrhythmia, uncontrolled congestive heart failure, third degree heart block, pericarditis, myocarditis, pulmonary/systemic embolism within the past 6 months, thrombophlebitis, ST displacement > 3 mm at rest, history of cardiac arrest)
* Contraindications for exercise testing118 including: recent (within 6 months) cardiac event (MI, pulmonary edema, myocarditis, pericarditis), unstable angina, uncontrolled arrhythmia, third degree heart block, left bundle branch block, acute congestive failure, recent (within 6 months) pulmonary/systemic embolus, severe electrolyte abnormality
* Meets criteria to stop screening exercise test118 as decided by overseeing physician (Dr. Schwartz or McTiernan)
* volunteering in order to lose weight
* alcohol or drug abuse, significant mental illness (as assessed by study staff impression)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 1997-01; Primary Completion 2003-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Serum total estrone concentration | Baseline, 3 month, 12-month

SECONDARY OUTCOMES:
serum total estradiol, free estradiol, estrone sulfate, testosterone, androstenedione, and sex hormone binding globulin (SHBG). | baseline, 3 month, 12-month
Urinary estrogen metabolite ratio (2-OHE1:16alpha-OHE1). | Basline, 3 month, 12-month
Adipose tissue stores: weight, body mass index, total fat mass, waist and hip circumferences and their ratio, and subcutaneous and intra-abdominal fat areas | Baseline, 3 month, 12 month
Fasting serum concentrations of insulin, glucose, and triglycerides | Baseline, 3 month, 12 month
Quality of life | Baseline, 3 month, 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Campbell PT, Wener MH, Sorensen B, Wood B, Chen-Levy Z, Potter JD, McTiernan A, Ulrich CM. Effect of exercise on in vitro immune function: a 12-month randomized, controlled trial among postmenopausal women. J Appl Physiol (1985). 2008 Jun;104(6):1648-55. doi: 10.1152/japplphysiol.01349.2007. Epub 2008 Apr 10. PMID 18403448
- [Result] Boynton A, Neuhouser ML, Sorensen B, McTiernan A, Ulrich CM. Predictors of diet quality among overweight and obese postmenopausal women. J Am Diet Assoc. 2008 Jan;108(1):125-30. doi: 10.1016/j.jada.2007.10.037. PMID 18155998
- [Result] Tworoger SS, Sorensen B, Chubak J, Irwin M, Stanczyk FZ, Ulrich CM, Potter J, McTiernan A. Effect of a 12-month randomized clinical trial of exercise on serum prolactin concentrations in postmenopausal women. Cancer Epidemiol Biomarkers Prev. 2007 May;16(5):895-9. doi: 10.1158/1055-9965.EPI-06-0701. PMID 17507612
- [Result] Rhew I, Yasui Y, Sorensen B, Ulrich CM, Neuhouser ML, Tworoger SS, Chubak J, Bowen DJ, McTiernan A. Effects of an exercise intervention on other health behaviors in overweight/obese post-menopausal women. Contemp Clin Trials. 2007 Jul;28(4):472-81. doi: 10.1016/j.cct.2007.01.002. Epub 2007 Jan 12. PMID 17287149
- [Result] Chubak J, McTiernan A, Sorensen B, Wener MH, Yasui Y, Velasquez M, Wood B, Rajan KB, Wetmore CM, Potter JD, Ulrich CM. Moderate-intensity exercise reduces the incidence of colds among postmenopausal women. Am J Med. 2006 Nov;119(11):937-42. doi: 10.1016/j.amjmed.2006.06.033. PMID 17071161
- [Result] Bowen DJ, Fesinmeyer MD, Yasui Y, Tworoger S, Ulrich CM, Irwin ML, Rudolph RE, LaCroix KL, Schwartz RR, McTiernan A. Randomized trial of exercise in sedentary middle aged women: effects on quality of life. Int J Behav Nutr Phys Act. 2006 Oct 4;3:34. doi: 10.1186/1479-5868-3-34. PMID 17020620
- [Result] Littman AJ, Vitiello MV, Foster-Schubert K, Ulrich CM, Tworoger SS, Potter JD, Weigle DS, McTiernan A. Sleep, ghrelin, leptin and changes in body weight during a 1-year moderate-intensity physical activity intervention. Int J Obes (Lond). 2007 Mar;31(3):466-75. doi: 10.1038/sj.ijo.0803438. Epub 2006 Aug 15. PMID 16909130
- [Result] Chubak J, Ulrich CM, Tworoger SS, Sorensen B, Yasui Y, Irwin ML, Stanczyk FZ, Potter JD, McTiernan A. Effect of exercise on bone mineral density and lean mass in postmenopausal women. Med Sci Sports Exerc. 2006 Jul;38(7):1236-44. doi: 10.1249/01.mss.0000227308.11278.d7. PMID 16826020
- [Result] Mohanka M, Irwin M, Heckbert SR, Yasui Y, Sorensen B, Chubak J, Tworoger SS, Ulrich CM, McTiernan A. Serum lipoproteins in overweight/obese postmenopausal women: a one-year exercise trial. Med Sci Sports Exerc. 2006 Feb;38(2):231-9. doi: 10.1249/01.mss.0000184584.95000.e4. PMID 16531889
- [Result] Chubak J, Tworoger SS, Yasui Y, Ulrich CM, Stanczyk FZ, McTiernan A. Associations between reproductive and menstrual factors and postmenopausal androgen concentrations. J Womens Health (Larchmt). 2005 Oct;14(8):704-12. doi: 10.1089/jwh.2005.14.704. PMID 16232102
- [Result] Frank LL, Sorensen BE, Yasui Y, Tworoger SS, Schwartz RS, Ulrich CM, Irwin ML, Rudolph RE, Rajan KB, Stanczyk F, Bowen D, Weigle DS, Potter JD, McTiernan A. Effects of exercise on metabolic risk variables in overweight postmenopausal women: a randomized clinical trial. Obes Res. 2005 Mar;13(3):615-25. doi: 10.1038/oby.2005.66. PMID 15833948
- [Result] McTiernan A, Sorensen B, Yasui Y, Tworoger SS, Ulrich CM, Irwin ML, Rudolph RE, Stanczyk FZ, Schwartz RS, Potter JD. No effect of exercise on insulin-like growth factor 1 and insulin-like growth factor binding protein 3 in postmenopausal women: a 12-month randomized clinical trial. Cancer Epidemiol Biomarkers Prev. 2005 Apr;14(4):1020-1. doi: 10.1158/1055-9965.EPI-04-0834. No abstract available. PMID 15824183
- [Result] Irwin ML, McTiernan A, Baumgartner RN, Baumgartner KB, Bernstein L, Gilliland FD, Ballard-Barbash R. Changes in body fat and weight after a breast cancer diagnosis: influence of demographic, prognostic, and lifestyle factors. J Clin Oncol. 2005 Feb 1;23(4):774-82. doi: 10.1200/JCO.2005.04.036. PMID 15681521
- [Result] Foster-Schubert KE, McTiernan A, Frayo RS, Schwartz RS, Rajan KB, Yasui Y, Tworoger SS, Cummings DE. Human plasma ghrelin levels increase during a one-year exercise program. J Clin Endocrinol Metab. 2005 Feb;90(2):820-5. doi: 10.1210/jc.2004-2081. Epub 2004 Dec 7. PMID 15585547
- [Result] Irwin ML, Tworoger SS, Yasui Y, Rajan B, McVarish L, LaCroix K, Ulrich CM, Bowen D, Schwartz RS, Potter JD, McTiernan A. Influence of demographic, physiologic, and psychosocial variables on adherence to a yearlong moderate-intensity exercise trial in postmenopausal women. Prev Med. 2004 Dec;39(6):1080-6. doi: 10.1016/j.ypmed.2004.04.017. PMID 15539040
- [Result] Chubak J, Tworoger SS, Yasui Y, Ulrich CM, Stanczyk FZ, McTiernan A. Associations between reproductive and menstrual factors and postmenopausal sex hormone concentrations. Cancer Epidemiol Biomarkers Prev. 2004 Aug;13(8):1296-301. PMID 15298949
- [Result] Frankenfeld CL, McTiernan A, Aiello EJ, Thomas WK, LaCroix K, Schramm J, Schwartz SM, Holt VL, Lampe JW. Mammographic density in relation to daidzein-metabolizing phenotypes in overweight, postmenopausal women. Cancer Epidemiol Biomarkers Prev. 2004 Jul;13(7):1156-62. PMID 15247126
- [Result] McTiernan A, Tworoger SS, Rajan KB, Yasui Y, Sorenson B, Ulrich CM, Chubak J, Stanczyk FZ, Bowen D, Irwin ML, Rudolph RE, Potter JD, Schwartz RS. Effect of exercise on serum androgens in postmenopausal women: a 12-month randomized clinical trial. Cancer Epidemiol Biomarkers Prev. 2004 Jul;13(7):1099-105. PMID 15247119
- [Result] Aiello EJ, Yasui Y, Tworoger SS, Ulrich CM, Irwin ML, Bowen D, Schwartz RS, Kumai C, Potter JD, McTiernan A. Effect of a yearlong, moderate-intensity exercise intervention on the occurrence and severity of menopause symptoms in postmenopausal women. Menopause. 2004 Jul-Aug;11(4):382-8. doi: 10.1097/01.gme.0000113932.56832.27. PMID 15243275
- [Result] Tworoger SS, Chubak J, Aiello EJ, Yasui Y, Ulrich CM, Farin FM, Stapleton PL, Irwin ML, Potter JD, Schwartz RS, McTiernan A. The effect of CYP19 and COMT polymorphisms on exercise-induced fat loss in postmenopausal women. Obes Res. 2004 Jun;12(6):972-81. doi: 10.1038/oby.2004.119. PMID 15229337
- [Result] Shade ED, Ulrich CM, Wener MH, Wood B, Yasui Y, Lacroix K, Potter JD, McTiernan A. Frequent intentional weight loss is associated with lower natural killer cell cytotoxicity in postmenopausal women: possible long-term immune effects. J Am Diet Assoc. 2004 Jun;104(6):903-12. doi: 10.1016/j.jada.2004.03.018. PMID 15175588
- [Result] Atkinson C, Lampe JW, Tworoger SS, Ulrich CM, Bowen D, Irwin ML, Schwartz RS, Rajan BK, Yasui Y, Potter JD, McTiernan A. Effects of a moderate intensity exercise intervention on estrogen metabolism in postmenopausal women. Cancer Epidemiol Biomarkers Prev. 2004 May;13(5):868-74. PMID 15159321
- [Result] McTiernan A, Tworoger SS, Ulrich CM, Yasui Y, Irwin ML, Rajan KB, Sorensen B, Rudolph RE, Bowen D, Stanczyk FZ, Potter JD, Schwartz RS. Effect of exercise on serum estrogens in postmenopausal women: a 12-month randomized clinical trial. Cancer Res. 2004 Apr 15;64(8):2923-8. doi: 10.1158/0008-5472.can-03-3393. PMID 15087413
- [Result] Tworoger SS, Yasui Y, Vitiello MV, Schwartz RS, Ulrich CM, Aiello EJ, Irwin ML, Bowen D, Potter JD, McTiernan A. Effects of a yearlong moderate-intensity exercise and a stretching intervention on sleep quality in postmenopausal women. Sleep. 2003 Nov 1;26(7):830-6. doi: 10.1093/sleep/26.7.830. PMID 14655916
- [Result] Irwin ML, Yasui Y, Ulrich CM, Bowen D, Rudolph RE, Schwartz RS, Yukawa M, Aiello E, Potter JD, McTiernan A. Effect of exercise on total and intra-abdominal body fat in postmenopausal women: a randomized controlled trial. JAMA. 2003 Jan 15;289(3):323-30. doi: 10.1001/jama.289.3.323. PMID 12525233
- [Derived] Duggan C, Xiao L, Wang CY, McTiernan A. Effect of a 12-month exercise intervention on serum biomarkers of angiogenesis in postmenopausal women: a randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2014 Apr;23(4):648-57. doi: 10.1158/1055-9965.EPI-13-1155. Epub 2014 Feb 5. PMID 24501378